CLINICAL TRIAL: NCT05619094
Title: The Effectiveness of Corrective Exercise Program on Alignment, Muscle Activation and Biomechanical Properties in Medical Students With Forward Head Posture
Brief Title: Effects of Exercise on Alignment and Muscle Parameters in Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Sibel Basaran, Head of Physical Medicine and Rehabilitation, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Cukurova125
Record Dates: First submitted 2022-10-27; First posted 2022-11-16 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Forward Head Posture
Keywords: Exercise; Craniovertebral angle; Muscle activation; Biomechanical properties; Surface electromyography
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corrective Exercise (Experimental): Selective corrective exercise program, 8 weeks
  Interventions: Other: Corrective exercise program
- Control (No Intervention): Training for proper posture

INTERVENTIONS:
Other: Corrective exercise program — Strengthening exercises for deep cervical flexor muscles and shoulder retractors.
  Stretching exercises for cervical extensors and pectoral muscles.
  Arms: Corrective Exercise

SUMMARY:
It is aimed to investigate the effect of corrective exercise program on alignment, muscle activation and biomechanical properties of muscles in medical students with forward head posture.

DETAILED DESCRIPTION:
Forward head posture (FHP) is a common postural abnormality that can be seen in all age groups. It is characterized by the head position being forward relative to the neck in the sagittal plane. The anterior displacement of the head is mainly assessed through examination of the craniovertebral angle (CVA) and a CVA of ˂50° is described as a FHP. Therapeutic exercises have shown to be effective in FHP and related symptoms in many studies. One of the exercise programs applied is the corrective exercise program. Within the scope of this program, deep cervical flexor muscles and shoulder retractors are strengthened, cervical extensors and pectoral muscles are stretched. This exercise protocol has been reported to provide relief in neck pain, improvement in CVA and shoulder angle. However, the number of studies examining the effect of corrective exercise program for the affected muscle groups in FHP on muscle activation parameters is limited, and there is no study examining the effect on the biomechanical properties of the muscles.

In this study, it is aimed to investigate the effect of corrective exercise program on alignment, muscle activation and biomechanical properties of muscles in medical students with forward head posture.

ELIGIBILITY:
Inclusion Criteria:

* Medical students with a Craniovertebral angle ˂ 50°

Exclusion Criteria:

* History of chronic pain in cervical region
* Presence of spinal deformity and malalignment
* Disease, fracture or surgery affecting the spine-shoulder-pelvic region
* Presence of malignancy
* BMI outside the normal range
* Presence of medical condition that prevents participation in physical exercise program
* Presence of neuromuscular disease
* Involvement in regular and professional sports activities

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Craniovertebral angle | Day 0
  The angle between the line connecting the seventh cervical vertebra and the tragus of right ear, and the horizontal line.
  running in the sagittal place through the C7 process
Craniovertebral angle | Week 8
  The angle between the line connecting the seventh cervical vertebra and the tragus of right ear, and the horizontal line.
  running in the sagittal place through the C7 process

SECONDARY OUTCOMES:
Surface electromyography (EMG) amplitude (RMS) | Day 0
  The activity levels of trapezius, sternocleidomastoid and pectoralis muscles will be measured with a wireless EMG system (Delsys, Inc, Boston, MA). The electrodes will be positioned on the belly of the muscle. The signals will be amplified and band-pass filtered (20-450 Hz) before being record digitally at 2000 samples per second, and then the root mean square (RMS) will be calculated. To normalize individual muscle contraction levels, we will use maneuvers of voluntary contractions.
Surface electromyography (EMG) amplitude (RMS) | Week 8
  The activity levels of trapezius, sternocleidomastoid and pectoralis muscles will be measured with a wireless EMG system (Delsys, Inc, Boston, MA). The electrodes will be positioned on the belly of the muscle. The signals will be amplified and band-pass filtered (20-450 Hz) before being record digitally at 2000 samples per second, and then the root mean square (RMS) will be calculated. To normalize individual muscle contraction levels, we will use maneuvers of voluntary contractions.
Myotonometer measures (Muscle tone) | Day 0
  The state of tension and biomechanical properties will be measured with a hand-held device (MyotonPro®, Myoton AS, Tallinn, Estonia). MyotonPro® displays the muscle mechanical properties by analyzing the oscillations of the myofascial tissue in response to the 10 short (15 ms) impulses, at 0.56 Newton (N) force and frequency of 1Hertz (Hz) applied by the probe of the device.
  The superficial muscles (trapezius, sternocleidomastoid and pectoralis muscle) will be evaluated.
  The device measures (computes simultaneously) the following parameters: Oscillation frequency (Hz), dynamic stiffness (N/m) and logarithmic decrement.
  Oscillation Frequency [Hz]: Characterizes the tone (intrinsic tension) of a muscle in its passive or resting state.
Myotonometer measures (Muscle stiffness) | Day 0
  The state of tension and biomechanical properties will be measured with a hand-held device (MyotonPro®, Myoton AS, Tallinn, Estonia). MyotonPro® displays the muscle mechanical properties by analyzing the oscillations of the myofascial tissue in response to the 10 short (15 ms) impulses, at 0.56 N force and frequency of 1Hz applied by the probe of the device.
  The superficial muscles (trapezius, sternocleidomastoid and pectoralis muscle) will be evaluated.
  The device measures (computes simultaneously) the following parameters: Oscillation frequency (Hz), dynamic stiffness (N/m) and logarithmic decrement.
  Dynamic Stiffness [N/m]: Characterises the resistance to a contraction or to an external force that deforms its initial shape.
Myotonometer measures (Muscle elasticity) | Day 0
  The state of tension and biomechanical properties will be measured with a hand-held device (MyotonPro®, Myoton AS, Tallinn, Estonia). MyotonPro® displays the muscle mechanical properties by analyzing the oscillations of the myofascial tissue in response to the 10 short (15 ms) impulses, at 0.56 N force and frequency of 1Hz applied by the probe of the device.
  The superficial muscles (trapezius, sternocleidomastoid and pectoralis muscle) will be evaluated.
  The device measures (computes simultaneously) the following parameters: Oscillation frequency (Hz), dynamic stiffness (N/m) and logarithmic decrement.
  Logarithmic Decrement: Characterises elasticity.
Myotonometer measures (Muscle tone) | Week 8
  The state of tension and biomechanical properties will be measured with a hand-held device (MyotonPro®, Myoton AS, Tallinn, Estonia). MyotonPro® displays the muscle mechanical properties by analyzing the oscillations of the myofascial tissue in response to the 10 short (15 ms) impulses, at 0.56 N force and frequency of 1Hz applied by the probe of the device.
  The superficial muscles (trapezius, sternocleidomastoid and pectoralis muscle) will be evaluated.
  The device measures (computes simultaneously) the following parameters: Oscillation frequency (Hz), dynamic stiffness (N/m) and logarithmic decrement.
  Ossilation Frequency [Hz]: Characterises the tone (intrinsic tension) of a muscle in its passive or resting state.
Myotonometer measures (Muscle stiffness) | Week 8
  The state of tension and biomechanical properties will be measured with a hand-held device (MyotonPro®, Myoton AS, Tallinn, Estonia). MyotonPro® displays the muscle mechanical properties by analyzing the oscillations of the myofascial tissue in response to the 10 short (15 ms) impulses, at 0.56 N force and frequency of 1Hz applied by the probe of the device.
  The superficial muscles (trapezius, sternocleidomastoid and pectoralis muscle) will be evaluated.
  The device measures (computes simultaneously) the following parameters: Oscillation frequency (Hz), dynamic stiffness (N/m) and logarithmic decrement.
  Dynamic Stiffness [N/m]: Characterises the resistance to a contraction or to an external force that deforms its initial shape.
Myotonometer measures (Muscle elasticity) | Week 8
  The state of tension and biomechanical properties will be measured with a hand-held device (MyotonPro®, Myoton AS, Tallinn, Estonia). MyotonPro® displays the muscle mechanical properties by analyzing the oscillations of the myofascial tissue in response to the 10 short (15 ms) impulses, at 0.56 N and frequency of 1Hz applied by the probe of the device.
  The superficial muscles (trapezius, sternocleidomastoid and pectoralis muscle) will be evaluated.
  The device measures (computes simultaneously) the following parameters: Oscillation frequency (Hz), dynamic stiffness (N/m) and logarithmic decrement.
  Logarithmic Decrement: Characterises elasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Aylin Sariyildiz, MD, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No